CLINICAL TRIAL: NCT05773781
Title: A Randomised Controlled Trial Investigating the Use of PuraBond® (3-D Matrix) in Transoral Resections of Primary Oral or Oropharyngeal Mucosal Lesions
Brief Title: PuraBond® and Pain Following Resection of Oral or Oropharyngeal Mucosal Lesions
Acronym: PuraBond PROOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UoL001737
Record Dates: First submitted 2023-03-02; First posted 2023-03-17 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-11

CONDITIONS: Pain; Hemorrhage; Hemostatics; Oropharynx; Oral Cavity
MeSH Terms: conditions — Pain; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PuraBond® (Active Comparator): Surgery with PuraBond® application to surgical field.
  Interventions: Other: PuraBond
- No PuraBond® (No Intervention): Surgery without PuraBond® application to surgical field.

INTERVENTIONS:
Other: PuraBond — Application of PuraBond to surgical field
  Arms: PuraBond®

SUMMARY:
To evaluate the use of Purabond® in transoral resections of primary oral or oropharyngeal lesions for diagnostic and therapeutic procedures. Patients will be enrolled and randomised to either have PuraBond® applied to the surgical field or not intra operatively. The primary outcome measure will assess if this intervention significantly reduces acute pain during the 30 day post-operative period alongside other post-operative complication rates and recovery outcomes.

DETAILED DESCRIPTION:
PuraBond® PROOF is a prospective, single centre, parallel group randomised controlled trial. Transoral approaches in head and neck surgery have become more common given they offer a minimally invasive approach to surgery, thus removing the need for external incisions in the neck. Post operative pain and bleeding are clinically important factor that directly impact patient recovery. PuraBond® is haemostatic agent, classified as a CE marked class III medical device, that is applied to surgical fields and has been shown to be both safe to use and effective in reducing bleeding. This trial will look to investigate the impact of applying PuraBond® in oral cavity or oropharyngeal operations on post-operative pain outcomes. Patients undergoing a pre-determined set of operations in either the mouth or oropharynx will be randomised to either receive PuraBond® to the surgical field during the operation or not. This allocation will be random and both treatments are currently used as part of routine standard clinical practice. Participants will be asked to monitor and record their pain levels pre and post-operatively by marking their pain level on a continuous scale from 'no pain' to 'the worse possible pain' using the Visual Analogue Scale (VAS). Patients will be enrolled from a single tertiary university hospital trust in the United Kingdom (Liverpool University Hospitals Foundation Trust). Case notes of all patients will also be analysed and data on patient demographics and post operative outcomes collated. This will be the first trial to look at PuraBond® use in head and neck surgery with pain being the primary trial outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient and disease factors are deemed suitable for transoral surgery under general anaesthetic.
* Decision to treat with primary transoral resection or local excision biopsy.
* Written informed consent provided.
* Clinically suspected or histologically confirmed primary dysplasia or malignancy of the oral cavity or oropharynx OR histologically confirmed diagnosis of squamous cell carcinoma in a cervical lymph node of unknown primary.
* Patient considered fit for surgery.

Exclusion Criteria:

* Lesions undergoing incisional or punch biopsy only.
* Surgery with planned primary closure or local/ distant flap reconstruction.
* Inability to provide written informed consent.
* Medical contraindication to a general anaesthetic or to PuraBond® use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool University Hospitals Foundation Trust (LUHFT), Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghazal Asswad R, Constable J, Abdelrahman A, Banks P, Mellor Z, Jones TM, Shaw R, Davies K, Loh C, Jackson R, Schache A, Fleming JC. The effect of PuraBond(R) on postoperative pain following transoral resections of primary oral or oropharyngeal neoplastic mucosal lesions: A blinded randomised controlled study (PuraBond(R) PROOF). Eur J Surg Oncol. 2025 Oct;51(10):110322. doi: 10.1016/j.ejso.2025.110322. Epub 2025 Jul 11. PMID 40669355

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PuraBond® | No PuraBond®
Started | 36 | 37
Completed | 32 | 36
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PuraBond® | No PuraBond® | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Continuous [Mean (Full Range); unit: years] | 64 [28 to 79] | 64 [45 to 81] | 64 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 26 | 25 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 36 | 68
Smoking status [Count of Participants; unit: Participants]
  Never | 14 | 21 | 35
  Ex-smoker | 12 | 12 | 24
  Current | 6 | 3 | 9
Primary tumour site [Count of Participants; unit: Participants]
  Oral cavity | 9 | 12 | 21
  Oropharynx | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cumulative Pain on the Visual Analogue Scale (VAS) at Postoperative Week 1
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 3.27 (2.75) | 4.35 (2.90)

2. Primary Outcome: Change From Baseline in Cumulative Pain on the Visual Analogue Scale (VAS) at Postoperative Week 2
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 2.95 (2.67) | 3.91 (2.91)

3. Primary Outcome: Change From Baseline in Cumulative Pain on the Visual Analogue Scale (VAS) at Postoperative Day 30
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 2.56 (2.63) | 3.41 (2.99)

4. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 1
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 2.46 (2.97) | 3.30 (3.06)

5. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 2
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 2.98 (2.79) | 3.87 (2.97)

6. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 4
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 3.36 (2.53) | 4.06 (2.72)

7. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 7
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 3.15 (2.61) | 4.28 (2.76)

8. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 14
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 31 | 33
score on a scale | 1.38 (1.55) | 1.66 (1.88)

9. Primary Outcome: Change From Baseline in Pain on the Visual Analogue Scale (VAS) at Day 30
Description: Visual Analogue Scale (VAS) score from 0 (no pain) to 10 (worst pain)
Time Frame: Baseline and day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 30 | 31
score on a scale | 0.23 (0.65) | 0.26 (1.88)

10. Secondary Outcome: Readmission
Description: Number of patients requiring hospital readmission
Time Frame: Within 30 days post operatively
Reporting Status: Not Posted

11. Secondary Outcome: Primary Haemorrhage
Description: Number of patients with primary haemorrhage
Time Frame: Within 24 hours post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 32 | 36
Participants | 0 | 0

12. Secondary Outcome: Secondary Haemorrhage
Description: Number of patients with secondary haemorrhage
Time Frame: Day 1 to day 30 post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 32 | 36
Participants | 2 | 6

13. Secondary Outcome: LOS
Description: Length of stay in hospital
Time Frame: Within 30 days post operatively
Reporting Status: Not Posted

14. Secondary Outcome: Primary Return to Theatre
Description: Number of patients requiring return to operating room
Time Frame: 24 hours post operatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 32 | 36
Participants | 0 | 0

15. Secondary Outcome: Secondary Return to Theatre
Description: Number of patients requiring return to operating room
Time Frame: Day 1 to day 30 postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | PuraBond® | No PuraBond®
Number analyzed (Participants) | 32 | 36
Participants | 1 | 1

16. Secondary Outcome: Oral Feeding
Description: Time taken to normal dietary intake
Time Frame: Within 30 days post operatively
Reporting Status: Not Posted

17. Secondary Outcome: Analgesia Use
Description: Drug, dose, route and frequency of post-operative analgesia usage
Time Frame: Within 30 days post operatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | PuraBond® | No PuraBond®
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/32 | 3/36
Other Adverse Events (participants affected / at risk) | 6/32 | 7/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PuraBond® (N=32) | No PuraBond® (N=36)
Haemorrhage (Surgical and medical procedures) | 1 | 1 — Haemorrhage requiring return to theatre for arrest of bleeding.
Haemorrhage (Surgical and medical procedures) | 0 | 1 — Haemorrhage requiring hospital readmission.
Cerebral infarct (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PuraBond® (N=32) | No PuraBond® (N=36)
Haemorrhage (Injury, poisoning and procedural complications) | 1 | 4
Wound infection (Infections and infestations) | 2 | 0
Chest infection (Infections and infestations) | 3 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
First bite syndrome (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT05773781/Prot_SAP_000.pdf